CLINICAL TRIAL: NCT06016309
Title: The MS-CEBA Study: Determining Cognitive, Energetic, Behavioural and Affective (CEBA) Profiles in Multiple Sclerosis
Acronym: MS-CEBA
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: University of Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: NL2023.202315914
Record Dates: First submitted 2023-07-25; First posted 2023-08-29 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Phase 1: In Phase 1 of the study, we aim to include a minimum of 300 patients to identify how often which CEBA symptoms occur among pwMS and which symptoms cluster together, forming CEBA profiles. In addition, in Phase 1, an on age and education level matched group of 100 Healthy controls will be included to allow comparison of performance-based measures.
  In Phase 2 of the study, we aim to include a minimum of 100 patients, after approximately two years, to investigate whether we can replicate the results of Phase 1, validating the different CEBA profiles.
  Interventions: Other: There is no intervention.
- Retest Phase 1: After a year, a retest of around 50 patients will take place in order to determine whether CEBA symptoms are stable over time which is important information in deciding whether CEBA profiles can be used as a guide for further care.
  Interventions: Other: There is no intervention.

INTERVENTIONS:
Other: There is no intervention. — There is no intervention.

SUMMARY:
Multiple Sclerosis (MS) is an invalidating neurological disease known to cause physical symptoms, which usually are the main focus of treatment. However, non-physical, more neuropsychological, symptoms also frequently occur, concerning the Cognitive, Energetic, Behavioural and Affective (CEBA) domains. Symptoms in the CEBA domains are known to negatively affect societal participation, and thereby quality of life. Unfortunately, despite their negative consequences, CEBA symptoms are not always timely recognized in people with MS (pwMS). Moreover, despite the fact that there are various effective neuropsychological treatments available for neurological patients with these symptoms, most pwMS do not yet receive these treatments.

Although findings in group studies confirm that each of the CEBA domains can be affected in pwMS and correlations between symptoms regarding different CEBA domains have been found, there are large differences between individual pwMS with regard to which CEBA symptoms co-occur and which CEBA symptoms prevail. In order to optimize care for pwMS (e.g. timely referring patients to suiting neuropsychological treatment) there is need for a large scale study investigating over the whole range of CEBA symptoms how frequent these occur, whether and how symptoms co-occur, and thus if CEBA profiles can be identified. Identification of CEBA profiles can serve to quickly identify pwMS with neuropsychological problems in clinical practice, and provide an indication for possible neuropsychological treatment. If CEBA profiles are identified, it is considered likely that multiple CEBA symptoms will be prominent within a single CEBA profile. Here, subjective burden of pwMS can play an important role in determining which symptoms the main focus should be on in possible neuropsychological treatment.

Currently, a clear and standardized procedure with a feasible neuropsychological screening instrument quickly identifying and combining CEBA profile and subjective burden, providing a suitable indication for possible neuropsychological treatment, is lacking.

The aim of the present study is identifying CEBA profiles in pwMS and subsequently developing a feasible screening instrument allowing quick identification of CEBA profile and subjective burden of pwMS in clinical practice, providing a suitable indication for possible neuropsychological treatment. If needed, combining of or adjustments to existing neuropsychological treatments will be suggested in order meet the needs of pwMS with CEBA symptoms. All of this with the ultimate aim to improve societal participation, and accordingly quality of life, of pwMS.

ELIGIBILITY:
In order to be eligible to participate in this study, a patient must meet all of the following criteria:

Inclusion Criteria:

* Confirmed MS diagnosis (all subtypes);
* Age18-70;
* Adequate command of the Dutch language.

Exclusion Criteria:

* Not being able to participate in a short neuropsychological assessment (NPA) as judged by the MS clinician and/or investigator;
* Presence of any other neurological and/or major psychiatric condition.

The group of HC's will be matched to the patient group on age and education level.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with Multiple Sclerosis (pwMS).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2027-07-20 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognition | 6-48 months
  The main study parameter is CEBA profile, which is latent and thus needs to be derived from the scores on neuropsychological tests and questionnaires regarding the CEBA domains, using latent profile analysis.
  Neuropsychological instruments regarding the Cognitive domain:
  * Neuropsychological tests for information processing speed (Symbol Digit Modalities Test & Trail Making Test A)
  * Neuropsychological tests for attentive/executive control (Trail Making Test A + B & Letterfluency)
  * Neuropsychological tests for memory (15 Word Test & Digit Span Test of the Wechsler Adult Intelligence Scale)
Energy | 6-48 months
  The main study parameter is CEBA profile, which is latent and thus needs to be derived from the scores on neuropsychological tests and questionnaires regarding the CEBA domains, using latent profile analysis.
  Neuropsychological instrument regarding the Energetic domain:
  - Questionnaire for mental and physical fatigue (Dutch Multifactor Fatigue Scale)
Behaviour | 6-48 months
  The main study parameter is CEBA profile, which is latent and thus needs to be derived from the scores on neuropsychological tests and questionnaires regarding the CEBA domains, using latent profile analysis.
  Neuropsychological instruments regarding the Behavioural domain:
  * Neuropsychological test for social cognition (Facial Expressions of Emotion - Stimuli and Tests)
  * Subscales of a questionnaire for social cognitive symptoms (Dysexecutive Questionnaire - self and proxy)
Affect | 6-48 months
  The main study parameter is CEBA profile, which is latent and thus needs to be derived from the scores on neuropsychological tests and questionnaires regarding the CEBA domains, using latent profile analysis.
  Neuropsychological instrument regarding the Affective domain:
  - Questionnaire for anxiety and depression (Hospital Anxiety and Depression Scale)

SECONDARY OUTCOMES:
Level of societal participation | 6-48 months
  Level of societal participation will be derived from the score on a questionnaire called 'Impact on Participation and Autonomy (IPA)'
Subjective burden | 6-48 months
  Subjective burden will be obtained through conducting an anamnesis.
Demographic information | 6-48 months
  Demographic information will be derived from medical records and anamnesis.

CONTACTS AND LOCATIONS:
Overall Officials: Joke Spikman, Prof. Dr., Principal Investigator — Department of Neurology - Unit Neuropsychology of the University Medical Center Groningen (UMCG)
Locations (1):
- University Medical Center Groningen (UMCG), Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Reinhardt A, Rakers SE, Heersema DJ, Beenakker EAC, Meilof JF, Timmerman ME, Spikman JM. Protocol for the MS-CEBA study: an observational, prospective cohort study identifying Cognitive, Energetic, Behavioural and Affective (CEBA) profiles in Multiple Sclerosis to guide neuropsychological treatment choice. BMC Neurol. 2024 Jun 28;24(1):224. doi: 10.1186/s12883-024-03737-6. PMID 38943063